CLINICAL TRIAL: NCT00867620
Title: Development of a Non-Invasive DNA Methylation-Based Assay System for the Risk Assessment of Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yeong-Shiau Pu, Department of Urology / National Taiwan University Hospital
Other Study IDs: 200707055R
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — These biospecimens will be keep in low-temperature (-80 degree)and then genomic DNA will be extracted from blood/urine samples until the detection of DNA methylation profiles.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: case group: patients with urothelial carcinoma
- 2: control group: those without previous history of any malignancy

SUMMARY:
Bladder cancer ranks the ninth in worldwide cancer incidence. Approximate 90% of bladder cancer is the malignancy of urothelium tissues, the urothelial cancer (UC). The mortality of bladder cancer is mainly due to recurrence and metastasis. Unfortunately, the currently available cytology or cystoscopy examination is of limited value because of low sensitivity of early disease. New biomarkers as well as detection technology are thus required to improve early diagnosis. By the aid of quantitative methylation-specific PCR (QMSP), which allows detecting tumor-derived DNA from tissues and body fluids, DNA methylation-based assay is thus developing for early detection and prognosis.

The goal of this proposed project is to develop a panel of DNA-methylation based biomarkers for UC diagnosis, prognosis, and prediction of responses to therapy (especially the recurrence, invasion, survival, and responses to therapeutic agents). Although numerous studies have investigated the aberrant promoter hypermethylation in bladder cancers or UC, inconsistent results are observed. DNA hypermethylation determination may rely on not only the conditions of QMSP, but also the biopsy specimens of different race, environmental expose factors, and regional variation. We thus need to profile the DNA methylation pattern of UC patients in Taiwan to establish a panel of potential prediction biomarkers for local patients.

DETAILED DESCRIPTION:
In the recent years, technologies of genomics, expression analysis and proteomics have been brought to guide the study of risk assessment and early detection of cancers. This proposed study aims to develop a non-invasive DNA methylation-based assay system elucidating a panel of aberrantly hypermethylated genes from urothelial tumors and urine sediments, to improve the risk assessment of urothelial carcinoma; such as early diagnosis, prognosis, and prediction of response to therapeutic regimes. This proposal will establish several techniques to study the methylation status on gene promoter regions. Three tasks will be achieved in this study: (1) Profiling the aberrant DNA methylation in urothelial carcinoma and determining potential prediction biomarkers. (2) Establishing a non-invasive assay by detecting DNA hypermethylation status in exfoliated cells collected from void urine; (3) Mapping the DNA hypermethylation changes from normal to malignant urothelial tumors and studying the underlying mechanism. Through the collaboration of a genetic toxicologist (Te-Chang Lee, PhD, IBMS), a urologist (Yeong-Shiau Pu, MD/PhD, NTUH) and epidemiologists (Hung-Yi Chiou, PhD, Taipei Medical University), we will explore the risk biomarkers for urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* those with histopathological-confirmed urothelial carcinoma will be included.

Exclusion Criteria:

* those were younger than 40 years old or with previous history of any other cancers will be excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects from the Department of Urology of NTUH. Those with urothelial carcinoma(bladder, renal pelvis and ureter) will be recruited in this study period. After they signed the informed consent,we will ask them some questions through face-to-face interview and collect 6-8ml blood and 50c.c. urine. Then genomic DNA will be extracted from these biospecimens to perform a non-invasive DNA methylation-based assay.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2008-08; Study Completion 2010-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: HUNG-YI CHIOU, PhD, Principal Investigator — COLLEGE OF PUBLIC HEALTH, TAIPEI MEDICAL UNIVERSITY; Yeong-Shiau Pu, MD, Principal Investigator — Department of Urology, National Taiwan University Hospital; Te-Chang Lee, PhD, Principal Investigator — Institute of Biomedical Sciences, Academia Sinica